CLINICAL TRIAL: NCT05686759
Title: A Phase 3b Study to Investigate the Safety and Efficacy of Undiluted Intravenous Infusion of I.V.-Hepabig Inj. in Post-liver Transplant Patients
Brief Title: A Study to Investigate the Safety and Efficacy of Undiluted Intravenous Infusion of I.V.-Hepabig Inj.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GC Biopharma Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GC5103-003_UDIV_P3b01
Record Dates: First submitted 2022-12-02; First posted 2023-01-17 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Liver Transplantation; Hepatitis B Immunoglobulin; Liver Diseases
MeSH Terms: conditions — Hepatitis B; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Undiluted intravenous infusion of I.V.-Hepabig inj (Experimental): Undiluted intravenous infusion of I.V.-Hepabig inj 10,000 International Unit within approximately 30 minutes
  Interventions: Biological: Undiluted I.V.-Hepabig inj(GC5103)
- Diluted intravenous infusion of I.V.-Hepabig inj (Active Comparator): Diluted intravenous infusion of I.V.-Hepabig inj 10,000 International Unit into Dextrose 5% in water within approximately 1 hour
  Interventions: Biological: Diluted I.V.-Hepabig inj(GC5103)

INTERVENTIONS:
Biological: Undiluted I.V.-Hepabig inj(GC5103) — undiluted I.V.-Hepabig inj(GC5103) 10,000 International Unit
  Arms: Undiluted intravenous infusion of I.V.-Hepabig inj
Biological: Diluted I.V.-Hepabig inj(GC5103) — Diluted I.V.-Hepabig inj(GC5103) 10,000 International Unit
  Arms: Diluted intravenous infusion of I.V.-Hepabig inj

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of undiluted intravenous infusion of I.V.-Hepabig inj. in post-liver transplant patients

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 and <65 years at the time of signing the consent form
2. Subjects who had history of liver transplantation due to HBV-related end-stage liver disease such as cirrhosis, liver cancer and fulminant hepatic failure and received treatment for prevent hepatitis B recurrence
3. HBsAg(+) before liver transplantation
4. Subjects who have been received I.V.-Hepabig inj more than 3 times dose of 10,000International Unit/4weeks regimen

Exclusion Criteria:

1. Subject with history of anaphylaxis to any component of the investigational product
2. Pregnant or breast-feeding women
3. Deficiency of Immunoglobulin A
4. Clinically significant renal diseases (serum creatinine >2.0mg/dL, anuria, renal failure or on dialysis at screening)
5. Hemophilia
6. Co-infection with Hepatitis A Virus, Hepatitis C Virus, or Human Immunodeficiency Virus
7. Subject with history of malignancy within the last 5 years (excluding primary liver cancer)
8. Subject received estrogen or hormone replacement therapy within 3 months before screening
9. HBsAg or HBeAg or HBV DNA positive at screening
10. Anti HBs titer less than below criteria at screening <150 IU/L for subject whose HBeAg and HBV DNA were negative(-) before liver transplantation >500 IU/L for subject whose HBeAg or HBV DNA were positive(+) before liver transplantation
11. Subject with history of drug abuse
12. Participated in another clinical study within 30 days (relative to the last dose of investigational product) before screening
13. Subject who are determined disqualified to join clinical trials by investigator

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events occurred during clinical trials | during 20 weeks post first Investigational product administration
  Safety will be assessed throughout the study through clinical safety evaluations(Adverse events)

SECONDARY OUTCOMES:
Positive rate of Hepatitis B Surface Antigen(HBsAg) | Screening, 0, 4, 8, 12, 16, and 20 weeks
  Hepatitis B Surface Antigen(HBsAg) will be tested at every visit(V1~V7)
Hepatitis B Surface Antibody(Anti HBs) titer | Screening, 0, 4, 8, 12, 16, and 20 weeks
  Hepatitis B Surface Antibody(Anti HBs) titer will be tested at every visit(V1~V7)
Positive rate of Hepatitis B e Antigen(HBeAg) | Screening, 0, 4, 8, 12, 16, and 20 weeks
  Hepatitis B e Antigen(HBeAg) will be tested at every visit(V1~V7)
Positive rate of Hepatitis B Virus DNA(HBV DNA) | Screening, 0, 4, 8, 12, 16, and 20 weeks
  Hepatitis B Virus DNA(HBV DNA) will be tested at every visit(V1~V7)
Laboratory tests | Screening, 0, 4, 8, 12, 16, and 20 weeks
  Change from baseline in safety laboratory tests results (hematology,chemistry, urine) (each visit)
Vital signs | Screening, 0, 4, 8, 12, 16, and 20 weeks
  Change from baseline in vital sign (Blood Pressure, Pulse Rate, Body Temperature) (each visit)
Physical examination | Screening, 0, 4, 8, 12, 16, and 20 weeks
  Change from baseline in physical examination (Appearance, Skin, Head/Neck, Thorax/Lungs etc) (each visit)

CONTACTS AND LOCATIONS:
Locations (8):
- South Korea (8):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Ajou University Medical Center, Suwon, Gyeonggi-do
  - Asan Medical Center, Seoul, Seoul
  - Inje University Haeundae Paik Hospital, Busan
  - Chungnam National University Hospital, Daejeon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No